CLINICAL TRIAL: NCT07315256
Title: Combined Ultrasonographic Skin-to-Epiglottis Distance With Modified Mallampati Versus Modified Mallampati Score Alone in Predicting Difficult Laryngoscopy During Tracheal Intubation Under General Anesthesia: A Prospective, Randomized Double Blinded Controlled Study
Brief Title: Combined Ultrasonographic Skin-to-Epiglottis Distance With Modified Mallampati Versus Modified Mallampati Score Alone in Predicting Difficult Laryngoscopy During Tracheal Intubation Under General Anesthesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Abdullah Badawy Abdullah, Resident at Anesthesia and ICU Department, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Ultrasound in Intubation
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Ultrasonographic; Mallampati Score; Mallampati Score, Difficult Intubation, Videolaryngoscope; Tracheal Intubation
Keywords: Difficult Laryngoscopy; Tracheal Intubation; Modified Mallampati

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Mallampati Only (Active Comparator): Adult elective surgical patients will undergo standard preoperative airway assessment using the modified Mallampati score only. No airway ultrasound will be performed. An experienced anesthesiologist, blinded to all preoperative assessments, will perform direct laryngoscopy for tracheal intubation and record the Cormack-Lehane grade on first attempt.
  Interventions: Diagnostic Test: Clinical Airway Assessment With Modified Mallampati Score
- Mallampati Plus Ultrasound Skin-to-Epiglottis Distance (Experimental): Adult elective surgical patients will undergo standard preoperative airway assessment with the modified Mallampati score plus point-of-care airway ultrasound to measure the midline skin-to-epiglottis distance using a high-frequency linear probe at the thyrohyoid membrane. The measurement is non-invasive and does not change clinical management. An experienced anesthesiologist, blinded to both Mallampati and ultrasound results, will perform direct laryngoscopy for tracheal intubation and record the Cormack-Lehane grade on first attempt.
  Interventions: Diagnostic Test: Ultrasound-Guided Skin-to-Epiglottis Distance Measurement

INTERVENTIONS:
Diagnostic Test: Ultrasound-Guided Skin-to-Epiglottis Distance Measurement — Point-of-care airway ultrasound of the anterior neck using a high-frequency linear probe (10-13 MHz) placed transversely at the thyrohyoid membrane to measure the vertical skin-to-epiglottis distance in millimeters. The scan is performed preoperatively in supine neutral position, is non-invasive and painless, and does not alter anesthetic or airway management, which follow standard clinical practice. This measurement is combined with the modified Mallampati score in the experimental arm to predict difficult laryngoscopy (Cormack-Lehane grade 3-4).
  Arms: Mallampati Plus Ultrasound Skin-to-Epiglottis Distance
Diagnostic Test: Clinical Airway Assessment With Modified Mallampati Score — Standard preoperative bedside airway assessment using the modified Mallampati score without airway ultrasound; performed in the sitting position with mouth opening and maximal tongue protrusion, used routinely to anticipate difficulty of laryngoscopy.
  Arms: Modified Mallampati Only

SUMMARY:
This study will evaluate how well an ultrasound measurement of the distance from the skin to the epiglottis, when combined with the modified Mallampati score, can predict difficult laryngoscopy in adult patients undergoing elective surgery under general anesthesia. Adult patients scheduled for surgery requiring tracheal intubation will be randomly assigned to two assessment strategies before anesthesia: one group will have the usual bedside airway assessment with modified Mallampati alone, and the other group will have modified Mallampati plus a quick, painless ultrasound scan of the front of the neck to measure the skin-to-epiglottis distance. During intubation, the anesthesiologist, who is blinded to the preoperative assessments, will grade the laryngoscopic view using the Cormack-Lehane classification, and the investigators will compare how accurately each assessment approach predicts difficult laryngoscopy (grade 3-4). The study does not change how anesthesia or airway management is performed; ultrasound and clinical assessments are added solely for measurement and data collection, with minimal risk to participants and potential future benefits in improving airway risk stratification and patient safety.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blinded controlled study designed to evaluate whether combining preoperative ultrasonographic skin-to-epiglottis distance (SED) with the modified Mallampati score improves prediction of difficult laryngoscopy compared with the modified Mallampati score alone in adult elective surgical patients undergoing tracheal intubation under general anesthesia. Eligible patients will be randomly assigned to one of two groups: Group A will undergo standard preoperative airway assessment including modified Mallampati score only, while Group B will receive both modified Mallampati assessment and ultrasound measurement of SED using a standardized anterior neck scanning protocol in the preoperative area.

All patients will subsequently undergo direct laryngoscopy for tracheal intubation in the operating room, performed by an experienced anesthesiologist who is blinded to the preoperative airway assessment results; the Cormack-Lehane laryngoscopic view during the first intubation attempt will be recorded as the reference standard for defining difficult laryngoscopy (grade 3-4). Additional data collected will include age, sex, body mass index, relevant comorbidities, and type of surgery to allow adjustment for potential confounders. The primary endpoint is the diagnostic accuracy (area under the receiver operating characteristic curve) of SED plus modified Mallampati versus modified Mallampati alone for predicting difficult laryngoscopy. Secondary endpoints include the correlation of SED with Cormack-Lehane grade, sensitivity, specificity, and predictive values of each assessment strategy, and exploratory subgroup analyses in higher-risk patients such as those with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years.
* ASA physical status I-II.
* Scheduled for elective surgery under general anesthesia requiring tracheal intubation with direct laryngoscopy.
* Able to provide written informed consent.

Exclusion Criteria:

* Emergency surgery.
* Known or suspected difficult airway requiring planned alternative intubation technique (e.g., awake fiberoptic).
* History of significant upper airway pathology, neck mass, prior neck surgery, or radiation affecting airway anatomy.
* Limited mouth opening, cervical spine instability, or contraindication to standard sniffing position.
* Pregnancy.
* Refusal or inability to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of Ultrasonographic Skin-to-Epiglottis Distance plus Mallampati vs Mallampati alone for difficult laryngoscopy | From induction of anesthesia to completion of first direct laryngoscopy (intraoperative, approximately 10 minutes).
  Area under the receiver operating characteristic (ROC) curve (AUC) of the combined ultrasound skin-to-epiglottis distance plus modified Mallampati score compared with the AUC of the modified Mallampati score alone for predicting difficult laryngoscopy, defined as Cormack-Lehane grade 3-4 on first direct laryngoscopy attempt.

SECONDARY OUTCOMES:
Correlation between skin-to-epiglottis distance and Cormack-Lehane grade | From preoperative ultrasound assessment to completion of first direct laryngoscopy (same operative session, approximately 30 minutes).
  Pearson or Spearman correlation coefficient between the ultrasound-measured midline skin-to-epiglottis distance and the Cormack-Lehane laryngoscopic grade recorded on the first intubation attempt in all patients who undergo airway ultrasound.